CLINICAL TRIAL: NCT01609491
Title: Comparison of the Effects of Phenylephrine and Norepinephrine on Hemodynamics and Tissue Oxygenation in Patients Undergoing Ophthalmic Surgery
Brief Title: Phenylephrine Versus Norepinephrine in Ophthalmic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: PheNor-001
Record Dates: First submitted 2012-01-17; First posted 2012-06-01 (Estimated); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Bloodpressure
MeSH Terms: interventions — Phenylephrine; Norepinephrine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- phenylephrine (Active Comparator): If the mean arterial pressure drops below 20% of the baseline value and/or below 90 mmHg, a syringe pump with phenylephrine will be started. The anaesthetist will be blinded for the type of vasopressor. Concentrations phenylephrine (20 µg /ml) will be used in the syringes
  Interventions: Drug: phenylephrine
- norepinephrine (Active Comparator): If the mean arterial pressure drops below 20% of the baseline value and/or below 90 mmHg, a syringe pump with norepinephrine (depending on randomisation) will be started. The anaesthetist will be blinded for the type of vasopressor. Concentrations Norepinephrine (10 µg/ml) will be used in the syringes
  Interventions: Drug: norepinephrine

INTERVENTIONS:
Drug: phenylephrine — If the mean arterial pressure drops below 20% of the baseline value and/or below 90 mmHg, a syringe pump with phenylephrine or norepinephrine (depending on randomisation) will be started. The anaesthetist will be blinded for the type of vasopressor. Concentrations phenylephrine (20 µg /ml) of Norepinephrine (10 µg/ml) will be used in the syringes
  Arms: phenylephrine
Drug: norepinephrine — If the mean arterial pressure drops below 20% of the baseline value and/or below 90 mmHg, a syringe pump with norepinephrine (depending on randomisation) will be started. The anaesthetist will be blinded for the type of vasopressor. Concentrations Norepinephrine (10 µg/ml) will be used in the syringes
  Arms: norepinephrine

SUMMARY:
In ophthalmic surgery the specific anaesthesiological challenges necessitate the administration of a combination of relatively high doses of hypnotics and analgetics. In order to preserve adequate organ perfusion, there is often a need to administer pharmacological agents for haemodynamic support. Depending on the experience of the anaesthetist a continuous infusion of phenylephrine or norepinephrine is used. It is currently not known which of these agents has the most favorable haemodynamical profile.

Haemodynamic parameters (continuous blood pressure, cardiac index, stroke volume and systemic resistance), peripheral tissue oxygenation and cerebral tissue oxygenation will be monitored noninvasively using the Nexfin® , Inspectra®, and Foresight® and O2C® monitoring devices.

ELIGIBILITY:
Inclusion Criteria:

Patients requiring general anaesthesia for ophthalmic surgery.

* Age > 18 years and older
* Diabetes or cardiovascular disease or age >55 years

Exclusion Criteria:

* Patient refusal
* Patient < 18 years

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2012-01; Primary Completion 2012-06 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
the haemodynamical effects of norepinephrine and phenylephrine during ophthalmic surgery | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Alain Kalmar, Dr, Principal Investigator — Anesthesiology
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands